CLINICAL TRIAL: NCT06905782
Title: Prospective Single Blinded Randomized Control Trial on the Effectiveness of Using Large Language Model Artificial Intelligence Chatbot to Improve Boston Bowel Preparation Score (BBPS) for Colonoscopy Preparation
Brief Title: Artificial Intelligence (AI) Technology May Help Patients to Understand Bowel Preparation Better Before They go for Colonoscopy.This Study Attempts to Leverage AI Chatbot in Counselling Patients to Improve Bowel Cleanliness, Reduce Anxiety as Well as Increase Procedural Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Nabil Mohammad Azmi, General Surgeon & Lecturer, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: JEP-2025-035
Record Dates: First submitted 2025-03-15; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Screening; Colon Polyps and Adenomas; Bowel Preparation Quality; Artificial Intelligence (AI)
Keywords: colorectal cancer; colon polyp; colonoscopy; bowel preparation; Boston Bowel Preparation Score (BBPS); artificial intelligence; AIChatbot; large language model; patient satisfaction; cancer screening
MeSH Terms: conditions — Colonic Polyps; Adenoma; Colorectal Neoplasms; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Prospective, single-masked, randomized control trial
Who Masked: Care Provider
Masking Description: Endoscopist performing the colonoscopy will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence (AI) Chatbot (Experimental): Patient's who will be interacting with AI chatbot for bowel preparation counselling
  Interventions: Procedure: AI chatbot study arm; Procedure: Traditional counselling study arm
- Conventional counselling by healthcare workers (Other): Patients receiving conventional way of counselling for bowel preparation before colonoscopy
  Interventions: Procedure: AI chatbot study arm; Procedure: Traditional counselling study arm

INTERVENTIONS:
Procedure: AI chatbot study arm — Intervention arm will have to undergo bowel preparation using standard polyethylene glycol solution (Fortrans)
Procedure: Traditional counselling study arm — Intervention arm will have to undergo bowel preparation using standard polyethylene glycol solution (Fortrans)

SUMMARY:
Traditional pre-colonoscopy counselling requires significant time from healthcare workers to explain procedures, limiting efficiency and patient turnover. Inadequate bowel preparation exacerbates this issue, leading to repeat procedures and increased costs. However, no study has yet evaluated the effectiveness of AI in improving the Boston Bowel Preparation Scale (BBPS) for colonoscopy preparation. By addressing this gap, AI chatbots could provide personalized guidance, reduce healthcare worker burden, improve preparation quality, and enhance patient experience.This research attempts to evaluate the effectiveness of using Artificial intelligence (AI) chat bot to improve bowel preparation, anxiety level and patient's satisfaction among colonoscopy patients in Hospital Tuanku Muhriz (HCTM), compared to conventional instructions

ELIGIBILITY:
Inclusion Criteria:

* All scheduled colonoscopy with indication
* Adequate digital literacy
* Adequate language literacy with Malay and English language

Exclusion Criteria:

* Patients with memory impairment due to previous stroke, dementia or Alzheimer's disease
* Diagnosed with clinical anxiety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of artificial intelligence (AI) chat bot in improving bowel preparation among colonoscopy patients in Hospital Tuanku Mukhriz (HCTM), compared to conventional instructions | 1 year
  Patients in interventional arm will be receiving counselling via interaction with AI chatbot.Each interaction session were limited to 15 minutes maximum. The quality of bowel preparation will be graded by the masked endoscopists using Boston Bowel Preparation Score (BBPS). Each of the three colon segments (right, transverse and left) will be assigned scores (0 - 3) . 0 - unprepared colon while 3 indicates the best possible preparation.A total score will range from 0 to 9, where higher scores indicate better bowel preparation.

SECONDARY OUTCOMES:
To determine the effectiveness of AI chat bot in relieving anxiety among colonoscopy patients in HCTM, compared to conventional instructions. | 1 year
  Anxiety level for both arms will be measured before and after colonoscopy using the validated Depression Anxiety and Stress Scale 21 (Anxiety Scale). Is a self-reporting scale that measure the the anxiety.DASS interpretation ;Normal 0-7, Mild 8-9, Moderate 10-14, Severe 15-19 and Extremely severe 20+
To determine the effectiveness of AI chat bot in improving satisfaction among colonoscopy patients in HCTM, compared to conventional instructions. | 1 year
  Patients from both arms will be interviewed after colonoscopy using the validated Patient Satisfaction Questionnaire (PSQ).PSQ are a set of questionnaires that help researchers to understand patient experiences and identify areas of improvement.Patients will be evaluated on multiple domains- general satisfaction, technical quality, interpersonal aspect, clarity of communication,access to care and confidence in healthcare provider. Each domain will be given scores according to the Likert scale ranging from 1 to 5. 1 means very dissatisfied while 5 means very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Mohammad Azmi, Doctor of General Surgery, Principal Investigator — Faculty of Medicine, The National University of Malaysia
Locations (1):
- Faculty of Medicine, The National University of Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol , Informed Consent Form, Clinical Study Report upon considerable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: APRIL 2025 - FEBRUARY 2026

REFERENCES:
- [Derived] Mohammad Azmi N, Abdul Jalal MI, Mohd Ashar SH, Mohd Nazri MI, Jie Y, Ganeson N, Augustine JK, Qian YS. A prospective single-masked, non-inferiority, parallel-group randomized controlled trial of the efficacy of a ChatGPT-based AI chatbot to improve Boston bowel preparation scores for colonoscopy preparation: A trial protocol. PLoS One. 2025 Oct 15;20(10):e0334349. doi: 10.1371/journal.pone.0334349. eCollection 2025. PMID 41091774

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT06905782/Prot_SAP_000.pdf